CLINICAL TRIAL: NCT03891173
Title: A Phase II, Open-Label, Randomized Study Immunoconjugate L-DOS47 in Combination With Vinorelbine/Cisplatin Versus Vinorelbine/Cisplatin Alone in Patients With Lung Adenocarcinoma
Brief Title: A Study of L-DOS47 in Combination With Vinorelbine/Cisplatin in Lung Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted at this time due to other budgetary priorities. Completion of reporting has been delayed first due to covid restrictions and more recently due to war in Ukraine.
Sponsor: Helix BioPharma Corporation (Industry)
Collaborators: KCR S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDOS003; 2016-003015-34 (EudraCT Number)
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Lung Adenocarcinoma
Keywords: lung adenocarcinoma; immunoconjugate; tumor microenvironment alkalinization
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Cisplatin; Vinorelbine

STUDY DESIGN:
Intervention Model Description: Part I includes a brief initial dose escalation phase, followed by Part II, which includes a randomized treatment phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- L-DOS47 in combination with cisplatin + vinorelbine (Experimental): L-DOS47 (6/9/12 µg/kg) is administered by iv on Day 1 and 8 of each 21-day treatment cycle, in combination with iv administration of standard cisplatin (80 mg/m2) on Day 2 + vinorelbine (30 mg/m2) on Day 2 and 9.
  Interventions: Drug: L-DOS47; Drug: Cisplatin; Drug: Vinorelbine
- Cisplatin + vinorelbine alone (Active Comparator): Administration by iv of standard Cisplatin (80 mg/m2) on Day 1 + vinorelbine (30 mg/m2) on Day 1 and 8 of each 21-day treatment cycle.
  Interventions: Drug: Cisplatin; Drug: Vinorelbine

INTERVENTIONS:
Drug: L-DOS47 — L-DOS47 lyophilized powder reconstituted and diluted for iv injection
  Arms: L-DOS47 in combination with cisplatin + vinorelbine
Drug: Cisplatin — Cisplatin concentrate for solution for iv infusion
Drug: Vinorelbine — Vinorelbine concentrate for solution for iv infusion
  Other Names: vinorelbine tartrate

SUMMARY:
This study will determine the highest dose of L-DOS47 that can be given in combination with vinorelbine/cisplatin, evaluate safety and tolerability of L-DOS47 when given in combination with vinorelbine/cisplatin, and assess how effective this combination is in treating patients with lung adenocarcinoma compared to patients who are given vinorelbine/cisplatin alone.

DETAILED DESCRIPTION:
The study is divided into two parts. In part I, the maximum tolerated dose of L-DOS47, when given in combination with vinorelbine/cisplatin, will be determined. Cohorts of 3 patients will be recruited into three dosing cohorts (6, 9 and 12 µg/kg). All patients at a given dose level must complete the first treatment cycle (3 week period) before escalation in subsequent patients can proceed. The decision for escalation to the next dose level will be made after the safety data have been reviewed by the Trial Steering Committee (TSC). If a patient in any cohort experiences a dose limiting toxicity, an additional 3 patients will be enrolled, for a maximum of up to 18 patients in this initial dose escalation part of the study.

In part II, after the maximum tolerated dose of L-DOS47 in combination with vinorelbine/cisplatin has been determined, a further 118 patients will be randomized (1:1) to receive L-DOS47 in combination with vinorelbine/cisplatin, or vinorelbine/cisplatin alone. Efficacy will be assessed by time to progression (time from first day of study drug administration to documented disease progression), response rate (proportion of patients with a best overall response of complete response and partial response using the Response Evaluation Criteria in Solid Tumours [RECIST] version 1.1 criteria), and overall survival (time from first day of study drug administration to death due to any cause). Monitoring will include radiological evaluations every second cycle. Safety and tolerability of L-DOS47 in combination will also continue to be evaluated.

For all patients, treatment will continue either until the patient experiences disease progression, unacceptable toxicity, the patient withdraws consent or has completed four treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years old
2. Histologically confirmed lung adenocarcinoma, classified as:

   * Chemotherapy-naive patients with metastatic lung adenocarcinoma for whom vinorelbine/cisplatin would be appropriate therapy;
   * metastatic recurrent lung adenocarcinoma following prior surgery, radiation and/or adjuvant chemotherapy at least 6 months ago, for whom vinorelbine/cisplatin would be appropriate therapy;
   * Staging assessed according to Tumor Node Metastases (TNM), 8th edition and based on computed tomography (CT) scan;
   * Grade 1 - 4 adenocarcinoma
3. No prior adjuvant chemotherapy within 6 months of the first treatment day if there is recurrent disease
4. At least a single measurable lesion in accordance with the RECIST v1.1 criteria
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0-1
6. A life expectancy of ≥ 3 months
7. Adequate organ function as determined by the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
   * Platelet count ≥ 100 × 10^9/L
   * Haemoglobin (HGB) ≥ 9 g/dL
   * Creatinine clearance ≥ 60 mL/min calculated using the Cockcroft-Gault Formula and serum creatinine ≤ 1.5 × the upper limit of normal (ULN)
   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 3 × ULN or < 5 × ULN if liver abnormalities are due to underlying malignancy
   * Total bilirubin ≤ 1.5 × ULN Note: Blood transfusions administered for the sole purpose of meeting the study inclusion criteria between the time informed consent is signed and first dose of L-DOS47 is administered are not allowed.
8. Able to understand the information provided to them and to give written informed consent before any study activities are conducted
9. Willing and able to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
10. Not pregnant and do not plan to become pregnant during the study. Females of childbearing potential must provide a negative pregnancy test within the Screening period (Day 21 to 0) and agree to use adequate non-hormonal contraception (which includes but is not limited to double barrier or sexual abstinence) during the study and for a period of 90 days following the last dose of study treatment. Male patients and their female partners of child-bearing potential must agree to each use an approved form of contraception during the study and for a period of 90 days following the last dose of study treatment.

Exclusion Criteria:

1. Pregnant or nursing mother
2. Prior history of other malignancies with the exception of non melanoma skin cancer
3. Patients with a known positive Epidermal Growth Factor Receptor (EGFR) mutation or whose tumour harbour an anaplastic lymphoma kinase (ALK) translocation
4. Active central nervous system metastasis and/or leptomeningeal disease (known or suspected); Patients with asymptomatic brain metastases are eligible if they had local therapy more than 1 month before enrolment
5. Evidence of active infection
6. Received treatment in another clinical study within the 30 days before commencing study drug and have not recovered from side effects of a study drug, except for alopecia
7. A serious uncontrolled medical condition
8. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or hepatitis C positive
9. Sustained QT interval corrected for heart rate (QTc) with Fridericia's correction > 450 msec at Screening, or a history of additional risk factors for Torsades de pointes (e.g., heart failure, hypokalaemia, family history of long QT syndrome)
10. Pre-existing peripheral neuropathy Grade ≥ 1 CTCAE
11. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent or compliance with the requirements of the protocol
12. Receiving chemotherapy during the 30 days before study treatment start; are receiving radiotherapy, targeted therapy, hormonal therapy, immunotherapy, major surgery or other study drugs during the 4 weeks before study treatment start, or have not recovered from all treatment related toxicities to Grade ≤ 1, except for alopecia. (Radiotherapy is allowed for the symptomatic treatment of bone metastases.)
13. Taking systemic steroids (other than inhalers or topical steroids) or other medication to suppress the immune system
14. Participating (or planning to participate) in any other clinical trial during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | Up to 12 weeks
  Time from first day of study drug administration to documentation of disease progression (including death due to progression)

SECONDARY OUTCOMES:
Objective response rate as measured using RECIST v. 1.1 | Up to 12 weeks
  Proportion of patients with a best overall response of complete response and partial response
Overall survival | Up to 12 weeks
  Time to death as defined as time from first day of study drug administration to death to to any cause
Safety and tolerability of L-DOS47 in combination with vinorelbine/cisplatin: Frequency of treatment emergence adverse events in patients | Up to 12 weeks
  Frequency of treatment emergent adverse events in patients

CONTACTS AND LOCATIONS:
Overall Officials: Cezary Szczylik, MD, Ph.D., Principal Investigator — Europejskie Centrum Zdrowia Otwock
Locations (4):
- Europejskie Centrum Zdrowia Otwock, Otwock, Poland
- Ukraine (3):
  - Dnipropetrovsk City Multi-field Clinical Hospital #4, Dnipro
  - Sumy Regional Clinical Oncological Centre, Sumy
  - Vinnytsya Regional Clinical Oncological Centre, Vinnytsia

IPD SHARING:
Plan to Share IPD: No